CLINICAL TRIAL: NCT04609267
Title: Interactive Voice-Based Administration of the PHQ-9
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Collaborators: Oral Roberts University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020039
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: This study will be a repeated measure, mixed methods design (i.e., it will contain both qualitative and quantitative components). Newly admitted patients will be asked to complete the questionnaires (i.e., PHQ-9 and the UEQ) at two different time points (i.e., Baseline and 1-month follow-up). In order to reduce or control for order effects, the procedure will be counterbalanced.
Masking Description: The study will be counterbalanced with no masking components
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paper Baseline (Experimental): Half of the participants will complete the PHQ-9 in the traditional paper format at their first appointment. At their second appointment 1-month later, they will complete the PHQ-9 on the Mirror device equipped with Amazon Alexa.
  Interventions: Diagnostic Test: PHQ-9 - Mirror format
- Mirror Baseline (Experimental): Half of the participants will complete the PHQ-9 on the Mirror device equipped with Amazon Alexa at their first appointment. At their second appointment 1-month later, they will will complete the PHQ-9 in the traditional paper format.
  Interventions: Diagnostic Test: PHQ-9 - Mirror format

INTERVENTIONS:
Diagnostic Test: PHQ-9 - Mirror format — The intervention we will be using is a new delivery system of the PHQ-9 using an Amazon Alexa equipped Mirror device. This Mirror device is similar to a smart television with a mirror interface. The device records auditory responses to the PHQ-9. We will be comparing the responses from the Mirror device to those given on the clinically established paper format.
  Other Names: PHQ-9 - Amazon Alexa equipped device

SUMMARY:
This study investigates a new delivery method for the Patient Health Questionnaire - 9 (PHQ-9), a clinically accepted tool for diagnosing major depressive disorder. The new tool records auditory responses to the assesment and the study will examine if the instrument is effective at capturing participant depression levels. If proven effective, future studies may investigate if the new format can be used to improve at home clinical care.

DETAILED DESCRIPTION:
This study is an investigation of a new delivery system of the Patient Health Questionnaire - 9 (PHQ-9), a clinically accepted tool for diagnosing major depressive disorder. The purpose of the study is to examine if the new delivery system of the PHQ-9 is effective at capturing participant depression levels. The new version uses a Mirror device, which is similar to a smart television with a mirror interface. The device records auditory responses to the PHQ-9 through Amazon Alexa. We will be comparing the responses from the Mirror device to those given on the clinically established paper format. If proven effective at capturing depression levels of patients, future studies may investigate if the new format can be used to improve at home clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Newly admitted patients to the Oklahoma State University Behavioral Medicine Clinic

Exclusion Criteria:

* Vulnerable populations, such as children (i.e., minors or individuals under the legal age of consent) and individuals who are incarcerated (i.e., prisoners), will be excluded.
* Individuals who are not their own guardian (i.e., those suffering from severe disabilities) will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-11-03 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
PHQ-9 Total Scores | Immediate
  Measure for Major Depressive Disorder from questionnaire responses
User Experience Survey | Immediate
  26 item questionnaire tracking user experience

CONTACTS AND LOCATIONS:
Overall Officials: Jason Beaman, D.O., Principal Investigator — Oklahoma State University Center for Health Sciences
Locations (1):
- OSU Behavioral Health Clinic, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data and findings will be posted on ClinicalTrials.gov.